CLINICAL TRIAL: NCT01200472
Title: A Phase 2, Multicenter, Randomized, Doubleblind, Placebo-controlled, Parallel-group,Efficacy Study of Apremilast (CC-10004)in Subjects With Erosive Hand Osteoarthritis
Brief Title: Efficacy Study of Apremilast (CC-10004) in Subjects With Erosive Hand Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACCOST Version 22-Oct-09; 2008-005365-61 (EudraCT Number)
Record Dates: First submitted 2010-04-08; First posted 2010-09-13 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Erosive Osteoarthritis of the Hand
Keywords: EHOA
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apremilast capsules (Experimental): Apremilast in 10 mg capsules
  Interventions: Drug: Apremilast
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — Apremilast is supplied as 10 mg capsules for oral administration. After a 7-day titration phase patients will receive 20 mg PO BID apremilast.
  Arms: Apremilast capsules
Drug: Placebo — Placebo capsules identical to apremilast
  Arms: Placebo

SUMMARY:
STUDY DESIGN:

This is a phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel-group, efficacy and safety study in 30 patients with erosive osteoarthritis of interphalangeal joints. The study is composed of 4 phases: a pre-randomization phase for up to 35 days followed by a 91-day randomized, double-blind two arm treatment phase, followed by a 77-day open label treatment phase for all study participants and a 28-day observational follow-up phase. Efficacy of the double blind and open label phase will be assessed at study day 84 and 168 after treatment start respectively.

STUDY DURATION:

The study length will be approximately 231 days for individual patients. With approximately a 12 month recruitment period the study is planned to last from January 2010 until July 2011 (19 months).

STUDY OBJECTIVES:

The primary objective is to evaluate the 84-day efficacy of apremilast 20 mg twice per day [BID], subsequent to a 7-day dose titration, compared with placebo, for the treatment of the symptoms of erosive hand osteoarthritis. Further objectives are to evaluate the effects on pain, disease activity, structural damage, quality of life, safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Must have at least two bone erosions detectable in conventional radiographs of the hands at the first carpo-metacarpal joint (CMC), proximal and/or distal interphalangeal joints
* Must have active disease at screening and randomization with at least two swollen and tender PIP and/or DIP joints; with the same two joints affected at both screening and randomization.
* Must have a patients self assessment of pain at baseline of at least 40% on a VAS
* Must have negative rheumatoid factor (RF) and anti-CCP antibody
* Must be able to adhere to the study visit schedule and other protocol requirements
* Male subjects (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in reproductive sexual activity with Females of Childbearing Potential (FCBP)while on study medication and for at least 28 days after taking the last dose of study medication
* Females of childbearing potential (FCBP) must have a negative urine pregnancy test at Screening and Baseline and must be willing to use one highly-effective form of birth control when engaging in reproductive sexual activity while on study medication and for at least 28 days after taking the last dose of study medication (§ A female of childbearing potential is a sexually mature female who 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been postmenopausal for at least 24 consecutive months (ie, has had menses at any time during the preceding 24 consecutive months).

Must meet the following laboratory criteria:

* Hemoglobin ≥ 9 g/dL
* Hematocrit ≥ 27%
* White blood cell (WBC) count ≥ 3000 /μL (≥ 3.0 X 109/L) and ≤ 14,000/μL (< 14 X 109/L)
* Platelets ≥ 100,000 /μL (≥ 100 X 109/L)
* Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L)
* Total bilirubin ≤ 2.0 mg/dL
* Aspartate transaminase (AST, SGOT]) and alanine transaminase(ALT, SGPT]) ≤ 1.5x upper limit of normal (ULN)

Exclusion criteria:

* History of any clinically significant cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic, or other major diseases
* History of any clinically significant inflammatory disease other than EHOA, especially, but not limited to, rheumatoid arthritis or spondylarthropathies
* History or Diagnosis of Fibromyalgia
* Evidence of gout, pseudogout or hemochromatosis
* Any injury, medical or surgical procedure to the affected joint(s) that may interfere with evaluation of the target hand OA joint(s)
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Pregnant or lactating female
* History of active Mycobacterium tuberculosis infection within 3 years prior to the screening visit. Infections that occurred > 3 years prior to entry must have been effectively treated
* History of incompletely treated latent Mycobacterium tuberculosis infection (as indicated by a positive Purified Protein Derivative [PPD] skin test or in vitro test (QuantiFERON Gold®).
* History of infected joint or joint prosthesis within the past 5 years
* Any anti-inflammatory or immunosuppressive therapy for any condition including, but not limited to, glucocorticoids, methotrexate, sulfasalazine, leflunomide, chloroquine, hydroxychloroquine, gold compounds, parenteral corticosteroids, penicillamine, cyclosporine, oral retinoids, mycophenolate mofetil, thioguanine, hydroxyurea, sirolimus, tacrolimus and azathioprine within 35 days of randomization and throughout the study
* Use of NSAIDs within 35 days of randomization and throughout the study
* Intra-articular corticosteroids for the targeted joints within three months prior to randomization
* Intra-articular injection of hyaluronate for the targeted joints within six month prior to randomization
* Use of any investigational medication within 35 days prior to randomization or 5 half-lives if known (whichever is longer)
* Use of "nutraceuticals" and alternative medicine products, unless taken at a stable dose for a minimum of three month prior to randomization
* Any clinically significant abnormality on 12-lead ECG at screening as determined by the investigator
* History of malignancy within previous 5 years (except for treated basal-cell skin carcinoma and/or squamous-cell skin carcinoma)
* High-risk factor(s) for, or a history of, human immunodeficiency virus (HIV), hepatitis B, or hepatitis C virus infection
* Have a known history of serious infections (eg, hepatitis, pneumonia, or pyelonephritis) in the previous 3 months Have a history of alcohol or substance abuse within the preceding 6 months that, in the opinion of the investigator, may increase the risks associated with study participation or study agent administration, or may interfere with interpretation of results
* Have participated in this study before
* Patients who are underage or are incapable to understand the aim, importance and consequences of the study and to give legal informed consent (according to § 40 Abs. 4 and § 41 Abs. 2 und Abs. 3 AMG).
* Patients who possibly are dependent on the sponsor or investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08; Primary Completion 2013-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in each treatment group who achieve a significant 50% improvement in AUSCAN Index at day 84 after treatment start compared with baseline | Day 84 after treatment start compared with baseline
  Proportion of subjects in each treatment group who achieve a significant 50% improvement in AUSCAN Index at day 84 after treatment start compared with baseline.

SECONDARY OUTCOMES:
Absolute values and change from baseline of the Patient self Assessment score (VAS) from baseline, day 84 and day 168 as well as proportion of patients in each treatment group who achieve improvements | Day 84 and at day 168 after treatment start compared with Baseline
  Patients self assessment of pain (VAS)
Change of the Physicians and Patients self assessment of global status (VAS)score from baseline, day 84 and day 168. | Day 84 and at day 168 after treatment start compared with Baseline
  Physicians and Patients self assessment of global status (VAS)
Change of the HAQ score from baseline, day 84 and day 168 in each treatment group who achieve improvements | Day 84 and at day 168 after treatment start compared with Baseline
  HAQ
Change of the SACRAH score from baseline, day 84 and day 168 in each treatment group who achieve improvements | Day 84 and at day 168 after treatment start compared with Baseline
  SACRAH
Change of the duration of the joint stiffness from baseline, day 84 and day 168 in each treatment group who achieve improvements | Day 84 and at day 168 after treatment start compared with Baseline
  Duration of joint stiffness
Change of swollen and tender joints from baseline compared to day 84 and day 168 in each treatment group. | Day 84 and at day 168 after treatment start compared with Baseline
  Swollen and tender joint counts
Measuring radiology changes from baseline, day 84 and day 168 using the RAMRIS score in each treatment. | Day 84 and at day 168 after treatment start compared with Baseline
  RAMRIS scoring system
Changes of the SF36 from baseline, day 84 and day 168 in each treatment group. | Day 84 and at day 168 after treatment start compared with Baseline
  SF36

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schett, MD, Study Director — University Hospital Erlangen, Department of Internal Medicine 3, Rheumatology and Clinical Immunology
Locations (3):
- Germany (3):
  - Prof. G. Schett, University Hospital Erlangen, Erlangen, Bavaria
  - Prof. Ulf Müller-Ladner, Kerckhoff-Klinik, Bad Nauheim
  - Prof. Matthias Schneider, Universitätsklinikum Düsseldorf, Klinik für Endokrinologie, Diabetologie und Rheumatologie, Düsseldorf